CLINICAL TRIAL: NCT01354600
Title: Short-term Positive Energy Balance and Exercise on 24-hour Plasma Levels of Hunger and Satiety Hormones in Sedentary Lean and Obese Men and Women
Brief Title: Effects of Positive Energy Balance and Exercise on Appetite Hormones in Sedentary Men and Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: H-2009-0001
Record Dates: First submitted 2011-05-05; First posted 2011-05-17 (Estimated); Last update posted 2013-07-23 (Estimated); Status verified 2013-07

CONDITIONS: Appetite and General Nutritional Disorders
Keywords: Obesity; Appetite; Hormones; Exercise; Body Weight
MeSH Terms: conditions — Obesity; Motor Activity; Body Weight | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Energy Balance (Other)
  Interventions: Other: Exercise or Sedentary
- Positive Energy Balance (Other)
  Interventions: Other: Exercise or Sedentary

INTERVENTIONS:
Other: Exercise or Sedentary — Daily cycling exercise at 50% maximal aerobic fitness for a total of ~120 minutes/day or no daily exercise (sedentary)

SUMMARY:
The purpose of this research study is to examine the effects of overfeeding and exercise on blood levels of hormones associated with regulating appetite, also thought of as feelings of hunger and satiety (fullness). Previous studies have shown that non-obese people have different amounts of these hormones in their blood compared to obese people.

The investigators hypothesize that exercise will promote improved insulin sensitivity and corresponding beneficial changes in obese individuals. The investigators predict exercise induced changes in 24-hour plasma hormone levels will be associated with improved appetite during overfeeding in obese individuals.

DETAILED DESCRIPTION:
In a randomized cross-over design, participants will complete two separate six-day & seven night inpatient stays (separated by at least 4 weeks) at the University of Wisconsin Hospital's Clinical and Translational Research Core (CTRC). During each six-day & seven night visit, participants will be fed an energy balance diet (energy intake = energy expenditure) for the first three days followed by three days of overfeeding (130% of the energy balance diet). During one of the inpatient periods, participants will exercise twice daily (once in the morning, once in the evening) for a total of approximately 120 minutes per day on an indoor exercise bicycle at ~50% of maximal aerobic fitness. During the other inpatient visit, participants will not exercise and will be inactive.

The investigators will examine the effect of short-term positive energy balance and exercise on 24-hour plasma levels of hormones related to hunger and satiety. These hormones include leptin, ghrelin, insulin, and peptide YY in sedentary lean and obese men and women. Our primary hypothesis is that when an obese person exercises, average 24-hour plasma leptin levels will increase in obese individuals during overfeeding compared to energy balance feeding, but fail to do so under sedentary conditions. In contrast, the investigators predict lean individuals will have an appropriate increase in average 24-hour leptin levels in response to overfeeding regardless of exercise treatment. Thus, the investigators suggest that a failure in the average 24-hour leptin response to overfeeding sets an obese person up for continued slow weight gain, as the leptin hunger signal fails to detect short-term overfeeding and does not produce a response. The investigators hypothesize that exercise will promote improved insulin sensitivity and increased leptin in the obese. The investigators predict that changes in average 24-hour plasma leptin levels will correlate with self-selected energy intake in lean individuals, but only during overfeeding plus exercise in obese individuals.

In addition, because the hunger and satiety response in humans is complex, this study will characterize the average 24-hour plasma levels of ghrelin, which stimulates hunger, and peptide YY, which stimulate satiety or fullness, in lean and obese individuals to determine if plasma levels are altered in obesity and in response to short-term positive energy balance.

Lastly, this study involves the banking of blood tissue specimens for future research. If it is decided such analysis is of scientific value, genetic analysis will be conducted for alterations in genes involved in the synthesis of, or receptors for, hunger and satiety hormones to be investigated under this study design.

ELIGIBILITY:
Inclusion Criteria:

* Healthy body mass index (BMI) = 19 < 25 kg/m2
* Obese BMI = 30 < 35 kg/m2
* Activity level = sedentary: Total energy expenditure/resting metabolic rate < 1.6 (average US adult level)

Exclusion Criteria:

* Tobacco use
* Regular exercise or physical activity, defined as > 2h/week of moderate to vigorous activity;
* Individuals who do not eat breakfast
* Weight loss of > 3% of body weight over the previous six months
* Eating a special diet (e.g., vegetarian or low-carbohydrate)
* Current diagnosis of, or using prescription medications for, thyroid dysfunction, type I or type II diabetes, hypertension, cardiovascular, kidney, or liver disease;
* Taking other prescription medications or over-the-country products that alter energy metabolism (other than birth control pills)
* Allergies to any of the foods used in the study
* Individuals who donated blood within 8 weeks prior to enrollment or who plan to give blood during the course of the study
* Claustrophobia
* History of exercise intolerance, including diagnosed exercise induced asthma or any physical limitations to seated cycling aerobic exercise
* Blood chemistries in excess of 130% of the upper normal level and/or hemoglobin or hematocrit below the normal range.
* Females that are pregnant (pregnancy status to be tested at the beginning of each 6-day metabolic chamber stay), lactating, or have irregular menses

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2009-05; Primary Completion 2011-11 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Blood plasma appetite hormone concentrations | Two separate six day & seven night inpatient visits, separated by at least 4 weeks.
  Blood samples will be drawn over 24 hours on the third and sixth day of each inpatient visit.

SECONDARY OUTCOMES:
Perceived subjective appetite measured by visual analog scales | Two separate six day & seven night inpatient visits, separated by at least 4 weeks.
  Appetite questionnaires will be filled out hourly as well as every 30 minutes after meals from 8:00am to 11:00pm on the third and sixth day of each inpatient visit.
Energy intake at a breakfast buffet | Two separate six day inpatient visits, separated by at least 4 weeks.
  A breakfast buffet will be served the morning after day 3 and day 6 of each inpatient visit to assess food intake following either energy balance (days 1-3) or overfeeding (days 4-6) with or without daily exercise.

CONTACTS AND LOCATIONS:
Overall Officials: Dale A Schoeller, PhD, Principal Investigator — University of Wisconsin-Madison, Dept. of Nutritional Sciences
Locations (1):
- University of Wisconsin Hospitals, Clinical and Translational Research Core (CTRC), Madison, Wisconsin, United States